CLINICAL TRIAL: NCT04168658
Title: A Pilot and Feasibility Cluster Randomized Controlled Trial of Physical Activity Program for Female Nursing Home Residents at Risk of Osteoporosis
Brief Title: A Physical Activity Program for Female Nursing Home Residents at Risk of Osteoporosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chengdu Jinjiang Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Li Tang, Assistant Professor, Chengdu Jinjiang Maternity and Child Health Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201909
Record Dates: First submitted 2019-11-16; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Chinese women; nursing home; physical activity; RCT
MeSH Terms: conditions — Osteoporosis; Motor Activity | interventions — Exercise; Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity and education intervention (Experimental)
  Interventions: Combination Product: Physical activity and education intervention
- Education intervention (Active Comparator)
  Interventions: Behavioral: Education intervention

INTERVENTIONS:
Combination Product: Physical activity and education intervention — At least six staff from each nursing home that assigned to the intervention group will be invited to attend two educational workshops. Participants in the intervention group will receive the following interventions.
  1. Face-to-face workshops: Five 1-hour educational workshops on physical activity will be delivered in months 1, 3, 5, 7 and 9 of the program held at each nursing home.
  2. Booklet: At the first educational workshop, each participant will be provided with a pictorial booklet.
  3. Exercise: The physical activity training consists of 50-60 min exercise sessions three times a week on non-consecutive days for 12 months.
  4. Others (newsletters, phone calls, and reminders): The intervention group will also receive newsletters containing myth dispelling information on osteoporosis and physical activity, motivational phone calls and a total of 52 SMS via mobile phones (reminders to attend workshop sessions and physical activity motivating messages) over 12 months.
  Arms: Physical activity and education intervention
Behavioral: Education intervention — Participants in the control group will only receive educational materials (i.e. face-to-face workshops and booklet) and will be wait listed to receive no other interventions of this study until after the post-intervention.
  Arms: Education intervention

SUMMARY:
Worldwide, osteoporosis causes more than 8.9 million fractures per annum. Osteoporosis used to be a significant public health concern that most commonly affected Caucasian women in Northern Europe and the United States. Recently, it has become a major public health problem in Asia, most notably among Chinese women.

We intend to conduct a cluster randomized controlled trial (RCT) to examine if a physical activity and education intervention, compared with an education-only intervention (waiting list for physical activity), can result in improved physical activity, reduced falls, and maintaining bone mass, among female nursing home residents in China. The aim of the current pilot and feasibility trial is to test the feasibility and acceptability of conducting these interventions.

A pilot and feasibility cluster RCT will be conducted for females aged 60 to 75 years living in nursing homes in Chengdu, the capital of Sichuan Province, Western China. The unit of cluster randomization is the nursing home. A total of four nursing homes (two state-owned and two private-owned) will be involved in the pilot and feasibility trial. They will be randomly selected and afterwards randomly assigned to either the intervention group (2 nursing homes) or control group (2 nursing homes). We seek to recruit 20 women from each nursing home.

The intervention group participants will exercise with the research staff or under supervision of the trained nursing home staff, and will receive face-to-face workshops, booklet, newsletters, phone calls, and short message service (SMS) reminders. Participants in the control group will only receive educational materials (i.e. face-to-face workshops and booklet) and will be wait listed to receive no other interventions of this study until after the post-intervention. All participants will be referred to doctors for advice and standard care as usual.

The primary outcome is the change of habitual physical activity from baseline to 12 months, which will be measured using the International Physical Activity Questionnaire - Short Form (IPAQ-SF). Secondary outcomes include incidental falls and change in bone mineral density (BMD) from baseline to 12 months. The study results will serve to provide an estimate of the effect size, intraclass correlation coefficient (ICC) and rates of eligibility, recruitment and attrition, which may enable a more accurate sample size calculation for a definitive RCT.

ELIGIBILITY:
Inclusion Criteria (cluster level-nursing home):

* have at least 100 female residents aged 60 to 75 years

Exclusion Criteria (cluster level-nursing home):

* are participating in any other clinical trials

Inclusion Criteria (participant level):

* female
* aged 60 to 75 years

Exclusion Criteria (participant level):

* have a previous diagnosis of osteoporosis
* are osteoporotic
* are taking medicines that would affect calcium or bone metabolism
* are already physically active (i.e. exercise at least three times a week at a moderate or higher intensity for ≥ 30 min)
* have taken part in any physical activity program within the past year
* sustain any medical condition that would put them at risk by taking part in moderate intensity exercises

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-02-10 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change of habitual physical activity | Baseline to 12 months post-baseline
  The primary outcome is the change of habitual physical activity from baseline to 12 months, which will be measured using the International Physical Activity Questionnaire - Short Form (IPAQ-SF).

SECONDARY OUTCOMES:
Incidental falls | 12 months starting from the baseline
  A fall is defined as "an event which results in a person coming to rest in advertently on the ground or floor or other lower level".
Change in bone mineral density (BMD) | Baseline to 12 months post-baseline
  BMD (g/cm2) of lumbar spine (L1-L4) and proximal femoral neck

CONTACTS AND LOCATIONS:
Overall Officials: Li Tang, PhD, Principal Investigator — Chengdu Jinjiang Maternity and Child Health Hospital